CLINICAL TRIAL: NCT03000114
Title: Comparison of Collagenase Injection and Percutaneous Needle Aponeurotomy for Treatment of Dupuytren's Disease
Brief Title: Collagenase Injection vs Percutaneous Needle Aponeurotomy for Dupuytren's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Justin Yeung, Doctor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB15-2463
Record Dates: First submitted 2016-12-17; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Dupuytren Contracture; Dupuytren's Disease of Finger
Keywords: Collagenase injection; percutaneous needle aponeurotomy
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Needle Aponeurotomy (Active Comparator): Percutaneous Needle Aponeurotomy (PNA) involves the surgeon anaesthetizing the skin over the Dupuytren's cord, then using a small gauge needle inserted percutaneously, cutting the cord with the sharp edge of the needle using a sweeping motion. This is repeated up the length of the cord to weaken it, allowing an extension force to be applied over the finger to rupture the cord.
  Interventions: Procedure: Percutaneous Needle Aponeurotomy
- Collagenase Injection (Active Comparator): Collagenase Injection (CI) involves the injection of collagenase clostridium histolyticum (0.58 mg), directly into the Dupuytren's cord. The patient then returns to see the surgeon within one week, has local anaesthetic is administered, and an extension force is applied to the affected digit to rupture the already weakened cord.
  Interventions: Drug: XIAFLEX

INTERVENTIONS:
Procedure: Percutaneous Needle Aponeurotomy
  Other Names: Percutaneous Needle Fasciotomy
  Arms: Percutaneous Needle Aponeurotomy
Drug: XIAFLEX
  Other Names: collagenase clostridium histolyticum
  Arms: Collagenase Injection

SUMMARY:
Dupuytren's disease is a non-curative, progressive disorder leading to function-impairing deformities of the hand. Although numerous treatments exist, the most common and widely accepted therapy is removal of diseased fascia. Surgery is limited by prolonged recovery time, and many patients require multiple surgeries throughout their life as the disease progresses, with repeat surgeries increasing the risk of complications.

Long recovery times and need for repeat surgeries has renewed interest in minimally invasive treatments for Dupuytren's disease. Percutaneous needle aponeurotomy (PNA) allows for rapid improvement in finger extension with minimal recovery time. The FDA approved collagenase clostridium histolyticum injection for Dupuytren's disease in 2010, which also allows for rapid increase in finger extension, also with minimal recovery time. Currently there is only one small study comparing PNA and collagenase injection (CI) that suggests similar outcomes in both treatments. Both treatments are minimally invasive, requiring minimal time off work and post-procedure pain. The main barrier to widespread adoption of CI is cost, particularly in patients with multiple areas of disease requiring treatment. The project proposed will compare these two methods for treating Dupuytren's disease.

Approximately 334 participants will be recruited from patients referred for treatment to hand surgeons trained in CI and PNA at two Calgary, AB hospitals. Need for treatment will be determined in the usual fashion, and the option for entry into the study will be proposed to patients meeting inclusion/exclusion criteria. Participants will be randomized into either the PNA or CI treatment group. The surgeon will not be blinded to the procedure group; however, the therapist measuring outcomes will be, and the study participants will need to not divulge to the therapists which group they are in.

Both procedures are performed under local freezing, and range from 5-20minutes. PNA involves the surgeon freezing the skin over the Dupuytren's cord, then using a small gauge needle inserted under the skin to cut the cord. This is repeated up the length of the cord to weaken it, allowing the surgeon to extend the finger and rupture the cord. CI involves the injection of collagenase (Xiaflex®), directly into the Dupuytren's cord. The patient then returns to see the surgeon within one week, has freezing placed in the hand, and the affected digit is extended to rupture the already weakened cord.

The patient will be required to present to the hand therapist team for measurements of joint angles before and after the assigned treatment is performed. In order to measure treatment efficacy, study participants will be required to return for measurements of treated joints every 6 months. Lastly, participants will need to inform the performing surgeon or therapist, at follow-up visits of any complications they experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring treatment for functionally limiting Dupuytren's disease involving the MCP and PIP joints, defined as MCP joint contracture 20-100 degrees, PIP joint contracture 20-80 degrees and positive table top test. Patients must be over 18 years of age to enroll in the study.

Exclusion Criteria:

* Patients who have had previous interventions of contracture presenting for treatment, in an effort to compare similar disease state and risk with each procedure.
* Disease involving DIP joint or thumb, as collagenase has not been approved for use in the thumb or DIP joints.
* Pregnant or nursing, although there is data indicating no detection of collagenase in patient serum following injection for Dupuytren's contractures, there is no data exploring the effects of collagenase on a fetus or infant.
* Anticoagulation therapy other than ASA (held 7 days prior to procedure), which is a recommendation by the manufacture of collagenase used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Contracture Recurrence | 6 months - 5 years
  Recurrence defined by an increase in joint contracture of at least 30 degrees in presence of palpable cord, or the patient underwent repeat intervention to correct new/worsening contracture in the treated joint.

SECONDARY OUTCOMES:
Patient Satisfaction | Intervention to 5 years post-intervention
  Survey
Complications | Intervention to 5 years post-intervention
  Patient to Report

CONTACTS AND LOCATIONS:
Overall Officials: Justin Yeung, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Desai SS, Hentz VR. The treatment of Dupuytren disease. J Hand Surg Am. 2011 May;36(5):936-42. doi: 10.1016/j.jhsa.2011.03.002. PMID 21527148
- [Background] Lermusiaux JL, Debeyre N. Le traitement médical de la maladie de Dupuytren. In: de Sèze S, Ryckewaert A, Kahn MF, Guérin CI. L'actualité rhumatologique 1979. Paris: Expansion Scientifique Française, 1980:338 -343.
- [Background] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771
- [Background] Gilpin D, Coleman S, Hall S, Houston A, Karrasch J, Jones N. Injectable collagenase Clostridium histolyticum: a new nonsurgical treatment for Dupuytren's disease. J Hand Surg Am. 2010 Dec;35(12):2027-38.e1. doi: 10.1016/j.jhsa.2010.08.007. PMID 21134613
- [Background] Nydick JA, Olliff BW, Garcia MJ, Hess AV, Stone JD. A comparison of percutaneous needle fasciotomy and collagenase injection for dupuytren disease. J Hand Surg Am. 2013 Dec;38(12):2377-80. doi: 10.1016/j.jhsa.2013.08.096. Epub 2013 Sep 20. PMID 24060510
- [Background] Chen NC, Shauver MJ, Chung KC. Cost-effectiveness of open partial fasciectomy, needle aponeurotomy, and collagenase injection for dupuytren contracture. J Hand Surg Am. 2011 Nov;36(11):1826-1834.e32. doi: 10.1016/j.jhsa.2011.08.004. Epub 2011 Oct 5. PMID 21981831
- [Background] Smith AC. Diagnosis and indications for surgical treatment. Hand Clin. 1991 Nov;7(4):635-42; discussion 643. PMID 1769986
- [Background] Peimer CA, Blazar P, Coleman S, Kaplan FT, Smith T, Lindau T. Dupuytren Contracture Recurrence Following Treatment With Collagenase Clostridium histolyticum (CORDLESS [Collagenase Option for Reduction of Dupuytren Long-Term Evaluation of Safety Study]): 5-Year Data. J Hand Surg Am. 2015 Aug;40(8):1597-605. doi: 10.1016/j.jhsa.2015.04.036. Epub 2015 Jun 18. PMID 26096221
- [Background] van Rijssen AL, Werker PM. Percutaneous needle fasciotomy in dupuytren's disease. J Hand Surg Br. 2006 Oct;31(5):498-501. doi: 10.1016/j.jhsb.2006.03.174. Epub 2006 Jun 12. PMID 16766101
- [Background] Zhang AY, Curtin CM, Hentz VR. Flexor tendon rupture after collagenase injection for Dupuytren contracture: case report. J Hand Surg Am. 2011 Aug;36(8):1323-5. doi: 10.1016/j.jhsa.2011.05.016. Epub 2011 Jun 25. PMID 21705158
- [Background] van Rijssen AL, Ter Linden H, Werker PMN. Five-year results of a randomized clinical trial on treatment in Dupuytren's disease: percutaneous needle fasciotomy versus limited fasciectomy. Plast Reconstr Surg. 2012 Feb;129(2):469-477. doi: 10.1097/PRS.0b013e31823aea95. PMID 21987045